CLINICAL TRIAL: NCT01735890
Title: A Randomized, Open-label, Single Dose, Two-way Crossover Clinical Trial to Compare the Safety, Pharmacokinetic Profiles of CJ Amlodipine/Valsartan 10/160mg Tablet and Novartis Exforge 10/160mg Tablet After a Single Oral Administration in Healthy Male Volunteers
Brief Title: Phase Ⅰ Study to Compare the Safety, Pharmacokinetic Profiles of CJ Amlodipine/Valsartan 10/160mg Tablet and Novartis Exforge 10/160mg Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ_AMV_102
Record Dates: First submitted 2012-11-25; First posted 2012-11-28 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: Safety; Pharmacokinetics
MeSH Terms: interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CJ Amlodipine/Valsartan 10/160mg (Experimental)
  Interventions: Drug: CJ Amlodipine/Valsartan 10/160mg Novartis Exforge 10/160mg
- Novartis Exforge 10/160mg (Active Comparator)
  Interventions: Drug: CJ Amlodipine/Valsartan 10/160mg Novartis Exforge 10/160mg

INTERVENTIONS:
Drug: CJ Amlodipine/Valsartan 10/160mg Novartis Exforge 10/160mg — single dose

SUMMARY:
The objectives of this study are:

* To compare the safety profile of CJ Amlodipine/Valsartan 10/160mg and Novartis Exforge 10/160mg after a single oral administration in healthy male volunteers
* To compare the pharmacokinetic profile of CJ Amlodipine/Valsartan 10/160mg and Novartis Exforge 10/160mg after a single oral administration in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Years 20-45
* 18 ≤ BMI < 27kg/m²
* volunteer

Exclusion Criteria:

* Subject taking inducer or inhibitor of drug metabolism enzyme such as barbital within 28days prior to study medication dosing
* Subject with symptoms of acute disease within 28days prior to study medication dosing
* Subject with gastrointestinal diseases or surgery which might significantly change absorption of medicines
* Use of any prescription medication within 14 days prior to study medication dosing and over-the-counter medication including oriental medication within 7 days prior to study medication dosing
* Subject with known for hypersensitivity reaction to amlodipine and valsartan
* Subject with any of the following conditions in laboratory test i. AST(sGOT) or ALT(sGPT) > Upper normal limit × 1.5 ii. Total bilirubin > Upper normal limit × 1.5 iii. eGFR< 50mL/min ⅳ. continued serum potassium concentration abnormal status (on baseline visit, < 3.5mEq/L or > 5.5mEq/L)
* Positive test results for HBs Ab, HCV Ab, Syphilis regain test
* Drug abuse or continued excessive use of caffeine (caffeine > five cups/day), severe heavy smoker (cigarette > 10 cigarettes per day) and alcohol(alcohol>30g/day)
* Subject who has been taken meal which affect on the absorption, distribution, metabolism, excretion of drug, especially grapefruit juice
* Clinically significant hypotension(SBP < 100mmHg, DBP ≤65mmHg) or hypertension(SBP 100mmHg, DBP < 65mmHg) when screening period
* Participation in any clinical investigation within 60days prior to study medication dosing
* Subjects with whole blood donation within 60days, component blood donation within 20days and blood transfusion within 30days prior to study medication dosing
* Subjects with decision of nonparticipation through investigator's review due to laboratory test results or other excuse such as non-responding to request or instruction by investigator

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic parameters of amlodipine and valsartan(Maximum plasma concentration (Cmax), Area under the plasma concentration curve (AUClast)) | Up to 144 hours

SECONDARY OUTCOMES:
AUCinf, Tmax, T1/2, CL/F | up to 144 hours

REFERENCES:
- [Derived] Nam JH, Oh M, Kim HJ, Han SK, Kim EJ, Song GS, Kim EY, Shin JG, Ghim JL, Kim HS. Pharmacokinetic comparison of amlodipine adipate/valsartan fixed-dose combination with amlodipine besylate/valsartan fixed-dose combination in healthy volunteers. Int J Clin Pharmacol Ther. 2015 Jan;53(1):66-74. doi: 10.5414/CP202045. PMID 25034618